CLINICAL TRIAL: NCT04706806
Title: Effect of Daily Vinegar Ingestion for Four Weeks on Mood State in Healthy College Students
Acronym: VIN2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00012406
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Mood; Depression
Keywords: acetic acid
MeSH Terms: conditions — Depression | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: randomized, controlled trial
Who Masked: Participant
Masking Description: Both groups received vinegar, either liquid form (active) or pill form (placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liquid vinegar (Experimental): 2 tablespoons (diluted in water) taken twice daily with meals
  Interventions: Dietary Supplement: apple cider vinegar
- vinegar pill (Placebo Comparator): 1 vinegar pill taken daily
  Interventions: Dietary Supplement: vinegar pill

INTERVENTIONS:
Dietary Supplement: apple cider vinegar — 2 tablespoons diluted in water taken twice daily with meals
  Other Names: apple cider vinegar (Bragg Live Food Products, LLC)
  Arms: liquid vinegar
Dietary Supplement: vinegar pill — one pill taken daily
  Other Names: Nature's Bounty Apple Cider Vinegar pills
  Arms: vinegar pill

SUMMARY:
The objective of this research is to record mood states and depression levels in healthy college students before and after 4 weeks of daily vinegar ingestion.

DETAILED DESCRIPTION:
Recent research suggests that fruit and vegetable intake is inversely associated with mood states and depression. Although the mechanism is not known, increased gut fermentation is suspected as changes in gut tryptophan metabolism was noted in these trials. Tryptophan is the precursor to serotonin, the neurotransmitter associated with improved mood state, but other metabolites of tryptophan have been associated with mental wellbeing as well. The main ingredient of vinegar, acetic acid, is the most common metabolite produced during gut fermentation of dietary fiber (mainly from fruits and vegetables) and can also be expected to influence the gut microbiome. It has been reported that vinegar ingestion is linked to a change in tryptophan metabolism in healthy adults consuming vinegar daily for 8 weeks. This study will explore the impact of vinegar ingestion on mood states.

ELIGIBILITY:
Inclusion Criteria:

* college student, non-athlete, no chronic health condition

Exclusion Criteria:

* vegetarians or others adhering to special diet, body mass index >30 kg/m2, pregnancy/lactation, unwilling to ingest vinegar

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
mood state | change from baseline at day 28
  Profile of Mood States (POMS) questionnaire score
depression | change from baseline at day 28
  Center for Epidemiologic Studies Depression Scale (CES-D)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No